CLINICAL TRIAL: NCT03474172
Title: Development and Validation of a Cloak Shape Device for Sham Pediatric Tuina
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou University of Traditional Chinese Medicine (Other)
Collaborators: Dongguan Kanghua Hospital (Other)
Responsible Party: Principal Investigator, Darong Wu, MD, PhD, Director,Program for Outcome Assessment in TCM, Professor, Chief Physician Affiliation: Guangzhou University of Traditional Chinese Medicine, Guangzhou University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: Z2017-212-01
Record Dates: First submitted 2018-03-06; First posted 2018-03-22 (Actual); Results first posted 2020-02-26 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Child
Keywords: Pediatric Tuina; Massage therapy; Sham Tuina; Sham massage; Sham device

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Genuine Tuina (Experimental): Participants will receive genuine tuina manipulated on their skin in addition to the conventional therapy given by the doctors. The whole process of the Tuina, which may last for 15 minutes, should be completed under the Cloak Shape device. After that the parents and the observers may be required to fill out corresponding questionnaires. The outcomes assessors will ask the child the sense perception of the manipulation via a questionnaire if he is equal or older than 3 years old.
  Interventions: Device: Cloak Shape Device for Genuine Tuina
- Sham Tuina (Sham Comparator): Except for the conventional therapy given by doctors, participants in this group will receive sham Tuina. A cloak shape device will be adopted, while inside the cover the therapist will use one hand to hold the childrens' hand or just put one hand on childrens' body and the other hand will do the manipulations on the therapist's own hand instead of childrens' hand or childrens' body. The acupoints and the manipulation time are the same as real Tuina group. Same questionnaires as those adopted in real Tuina group are also required to be completed.
  Interventions: Device: Cloak Shape Device for Sham Tuina

INTERVENTIONS:
Device: Cloak Shape Device for Sham Tuina — The Cloak Shape Device for Sham Tuina is exactly the same as the real one, which is opaque and big enough to cover the whole body and arms of a child who is under 6 years old. Two narrow holes are required on the cover, so that the therapist's hands can touch the child through these holes and a sham Tuina will be manipulated
  Arms: Sham Tuina
Device: Cloak Shape Device for Genuine Tuina — The Cloak Shape Device for Genuine Tuina is opaque and big enough to cover the whole body and arms of a child who is under 6 years old. Two narrow holes are required on the cover, so that the therapist's hands can touch the child through these holes and a genuine Tuina will be manipulated.
  Arms: Genuine Tuina

SUMMARY:
This study aims to evaluate the effectiveness of a Cloak Shape sham Pediatric Tuina device which can be applied in randomized controlled trials for Pediatric Tuina research.

DETAILED DESCRIPTION:
Chinese pediatric Tuina has been practiced as an option for health promotion, including disease prevention and treatment, more than one thousand years ago (652 AD). Many of the acupoints adopted in Chinese pediatric Tuina are located on children's fingers, hands and arms, which are unique if it is compared with those for adult tuina. The manipulation is found to be easily accepted by children, as the strength of tuina is gentle and soft. No severe adverse reaction in regards of Chinese pediatric Tuina was reported, the mild adverse reaction such as skin abrasion can be completely avoided with correct operating instructions. However, it is still lack of high quality RCTs (Randomized Controlled Trials) to evaluate its efficacy. The main obstacle is the difficulty to conduct a valid sham Tuina comparison group. In order to solve this problem, the investigators designed a device for sham Tuina, with a Cloak Shaped cover which is opaque and big enough to cover the whole body and arms of a child who is under 6 years old. Two narrow holes are required on the cover, so that the therapist's hands can touch the child through these holes. The whole manipulation process will be invisible under the cover.The investigators aim to detect whether it is effective as a sham device for pediatric Tuina researches.

ELIGIBILITY:
Inclusion Criteria:

1. Children with disease in Pediatric Outpatient Department of Kanghua Hospital
2. Children aged 0-6 years.
3. Guardian and child can be cooperative over the study period.
4. Guardian signed the informed consent.
5. Children have no attendance in other studies simultaneously.

Exclusion Criteria:

1. Child with one or more PT experiences on arms, abdomen or back.
2. Child with a previous history of convulsion.
3. Child with any of the following conditions on the area to be manipulated: phlebitis, open wound, fracture and tissue damage.
4. Child combined with any of following conditions: disorders of consciousness, seizures or twitching, shock, varicella, hand-foot-mouth disease, encephalitis B, and etc.

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2018-08-15 (Actual); Study Completion 2018-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darong Wu, MD,PhD, Principal Investigator — Guangzhou University of Traditional Chinese Medicine
Locations (1):
- Dongguan Kanghua Hospital, Dongguan, Guangdong, China

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All the recuitment work conducted at the outpatient department of pediatrics of Kanghua hospital where is a first class western medical hospital between May.2018 to August.2018.
Groups:
- Real Tuina: Children will receive real tuina manipulated on their skin in addition to the conventional therapy given by the doctors. The whole process of the Tuina, which may last for 15 minutes, should be completed under the Cloak Shape device. After that the parents and the observers may be required to fill out corresponding questionnaires. The outcomes assessors will ask the child the sense perception of the manipulation via a questionnaire if he is equal or older than 3 years old.
  Cloak Shape Device for Real Tuina: The Cloak Shape Device for Real Tuina is opaque and big enough to cover the whole body and arms of a child who is under 6 years old. Two narrow holes are required on the cover, so that the therapist's hands can touch the child through these holes and a real Tuina will be manipulated.
- Sham Tuina: Except for the conventional therapy given by doctors, children in this group will receive sham Tuina. A cloak shape device will be adopted, while inside the cover the therapist will use one hand to hold the childrens' hand or just put one hand on childrens' body and the other hand will do the manipulations on the therapist's own hand instead of childrens' hand or childrens' body. The acupoints and the manipulation time are the same as real Tuina group. Same questionnaires as those adopted in real Tuina group are also required to be completed by parents and observers.
  Cloak Shape Device for Sham Tuina: The Cloak Shape Device for Sham Tuina is exactly the same as the real one, which is opaque and big enough to cover the whole body and arms of a child who is under 6 years old. Two narrow holes are required on the cover, so that the therapist's hands can touch the child through these holes and a sham Tuina will be manipulated
Period: Overall Study
Arm/Group | Real Tuina | Sham Tuina
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This study enrolled children as the object to the Tuina therapy. As it is a study to assess the validation of blinding, the outcome assessment will mainly conduct among parents and observers . Questionaire will also be used for children who are over 3 yrs as they can understand. Therefore the units are child-parent-observer
Units Other Than Participants: child-parent-observer dyads
Groups:
- Sham Tuina: Except for the conventional therapy given by doctors, children in this group will receive sham Tuina. A cloak shape device will be adopted, while inside the cover the therapist will use one hand to hold the childrens' hand or just put one hand on childrens' body and the other hand will do the manipulations on the therapist's own hand instead of childrens' hand or childrens' body. The acupoints and the manipulation time are the same as real Tuina group. Same questionnaires as those adopted in real Tuina group are also required to be completed by parents, observers and children who are equal or older than 3 years old.
  Cloak Shape Device for Sham Tuina: The Cloak Shape Device for Sham Tuina is exactly the same as the real one, which is opaque and big enough to cover the whole body and arms of a child who is under 6 years old. Two narrow holes are required on the cover, so that the therapist's hands can touch the child through these holes and a sham Tuina will be manipulated
- Total: Total of all reporting groups
Arm/Group | Real Tuina | Sham Tuina | Total
Number analyzed (Participants) | 30 | 30 | 60
Number analyzed (child-parent-observer dyads) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: Month] — Age of 60 children
  Month | 14.76 (13.876) | 20.21 (18.849) | 17.98 (16.563)
Age, Continuous [Mean (Standard Deviation); unit: years] — Age of 60 parents
  years | 31.20 (4.473) | 32.07 (5.304) | 31.63 (5.002)
Sex: Female, Male [Count of Participants; unit: Participants] — Sex information of 60 children
  Participants
    Female | 13 | 10 | 23
    Male | 17 | 20 | 37
Sex: Female, Male [Count of Participants; unit: Participants] — Sex information of 60 parents
  Participants
    Female | 21 | 25 | 46
    Male | 9 | 5 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 30 | 30 | 60
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Education level of parents [Count of Participants; unit: Participants]
  Less than junior diploma | 5 | 2 | 7
  High school or junior college diploma | 18 | 20 | 38
  More than college diploma | 7 | 8 | 15
Occupation of parents [Count of Participants; unit: Participants]
  Professional person | 4 | 2 | 6
  Service personnel | 2 | 1 | 3
  Self-employed person | 1 | 4 | 5
  Laborer | 1 | 0 | 1
  Company stuff | 6 | 7 | 13
  Individual household or businessman | 6 | 6 | 12
  Housewife | 9 | 10 | 19
  Unemployed | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: The Accuracy Judgement Rates of the Type of Tuina That Children Received Based on Parents' Evaluations
Description: The accuracy judgement rate was calculated from the original data as below and was used as the primary outcome in the study.
Time Frame: The outcome measures started right after the PT therapy was completed and the measurement lasted for 10-15 mins.
Measure: Number; unit: parents
Groups:
- Real Tuina: Participants will receive real tuina manipulated on their skin in addition to the conventional therapy given by the doctors. The whole process of the Tuina, which may last for 15 minutes, should be completed under the Cloak Shape device. After that the parents and the observers may be required to fill out corresponding questionnaires. The outcomes assessors will ask the child the sense perception of the manipulation via a questionnaire if he is equal or older than 3 years old.
  Cloak Shape Device for Real Tuina: The Cloak Shape Device for Real Tuina is opaque and big enough to cover the whole body and arms of a child who is under 6 years old. Two narrow holes are required on the cover, so that the therapist's hands can touch the child through these holes and a real Tuina will be manipulated.
- Sham Tuina: Participants in this group will receive sham Tuina. A cloak shape device will be adopted, while inside the cover the therapist will use one hand to hold the childrens' hand or just put one hand on childrens' body and the other hand will do the manipulations on the therapist's own hand instead of childrens' hand or childrens' body. The acupoints and the manipulation time are the same as real Tuina group. Same questionnaires as those adopted in real Tuina group are also required to be completed.
  Cloak Shape Device for Sham Tuina: The Cloak Shape Device for Sham Tuina is exactly the same as the real one, which is opaque and big enough to cover the whole body and arms of a child who is under 6 years old. Two narrow holes are required on the cover, so that the therapist's hands can touch the child through these holes and a sham Tuina will be manipulated
Arm/Group | Real Tuina | Sham Tuina
Number analyzed (Participants) | 30 | 30
parents
  Parents who estimated the therapy is real Tuina | 28 | 25
  Parents who estimated the therapy is sham Tuina | 0 | 0
  Parents who were uncertain | 2 | 5

2. Primary Outcome: The Accuracy Judgement Rates of the Type of Tuina That Children Received Based on Observers' Evaluations
Description: as for outcome 1
Time Frame: The outcome measures started right after the PT therapy was completed and the measurement lasted for 10-15 mins.
Measure: Number; unit: observers
Arm/Group | Real Tuina | Sham Tuina
Number analyzed (Participants) | 30 | 30
observers
  Observers who estimated the therapy is real Tuina | 14 | 13
  Observers who estimated the therapy is sham Tuina | 3 | 7
  Observers who were uncertain | 13 | 10

3. Secondary Outcome: Verbal Rating Scale (VRS) of Parent's Attitude Towards Pediatric Tuina
Description: We adopt the VRS-4 to indicate diferent confident intensities towards pediatric Tuina from the perspective of parents as follow: not confident, somewhat confident, confident ,very confident.
Time Frame: The outcome measures started right after the PT therapy was completed and the measurement lasted for 10-15 mins.
Measure: Number; unit: parents
Arm/Group | Real Tuina | Sham Tuina
Number analyzed (Participants) | 30 | 30
parents
  Not confident | 0 | 1
  Somewhat confident | 17 | 17
  Confident | 10 | 11
  Very confident | 2 | 1

4. Secondary Outcome: Verbal Rating Scale (VRS) of Children's (≥3 Years Old) Perception of Pediatric Tuina
Description: We adopt the VRS-5 to indicate diferent discomfort intensities towards pediatric Tuina from the perspective of children equal or larger than 3 years old during and after the Tuina as follow: no discomfort; some discomfort; discomfort; very uncomfortable ; uncertain.
Time Frame: The outcome measures started right after the PT therapy was completed and the measurement lasted for 10-15 mins.
Measure: Number; unit: children
Arm/Group | Real Tuina | Sham Tuina
Number analyzed (Participants) | 7 | 3
children
  No discomfort | 7 | 3
  Some discomfort/discomfort/very uncomfortable | 0 | 0
  Uncertain | 0 | 0

5. Secondary Outcome: VRS of Parent's Attitude Towards Pediatric Tuina From the Observers' Perspectives
Description: We adopt the VRS-4 to indicate diferent trust intensities of the parents towards pediatric Tuina from the perspective of observers' perspectives as follow: Not confident, somewhat confident, confident, very confident.
Time Frame: The outcome measures started right after the PT therapy was completed and the measurement lasted for 10-15 mins.
Measure: Number; unit: parents
Arm/Group | Real Tuina | Sham Tuina
Number analyzed (Participants) | 30 | 30
parents
  Not confident | 0 | 0
  Somewhat confident | 15 | 18
  Confident | 12 | 9
  Very confident | 3 | 3

6. Secondary Outcome: Compliance of Guardians and Children for Three Continuous PT Therapies
Description: We adopt the VRS-4 to indicate diferent compliance intensities to follow 3 days continuous Tuina therapies as follow:improbable, somewhat improbable, probable, very probable.
Time Frame: The outcome measures started right after the PT therapy was completed and the measurement lasted for 10-15 mins.
Measure: Number; unit: parents
Arm/Group | Real Tuina | Sham Tuina
Number analyzed (Participants) | 30 | 30
parents
  Improbable | 0 | 0
  Somewhat improbable | 1 | 1
  Probable | 25 | 26
  Very probable | 4 | 3

ADVERSE EVENTS:
Time Frame: The adverse event data were collected during the Tuina therapy and 1 month after the therapy.
Groups:
- Sham Tuina: Except for the conventional therapy given by doctors, children in this group will receive sham Tuina. A cloak shape device will be adopted, while inside the cover the therapist will use one hand to hold the childrens' hand or just put one hand on childrens' body and the other hand will do the manipulations on the therapist's own hand instead of childrens' hand or childrens' body. The acupoints and the manipulation time are the same as real Tuina group. Same questionnaires as those adopted in real Tuina group are also required to be completed.
  Cloak Shape Device for Sham Tuina: The Cloak Shape Device for Sham Tuina is exactly the same as the real one, which is opaque and big enough to cover the whole body and arms of a child who is under 6 years old. Two narrow holes are required on the cover, so that the therapist's hands can touch the child through these holes and a sham Tuina will be manipulated
Arm/Group | Real Tuina | Sham Tuina
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-20): https://cdn.clinicaltrials.gov/large-docs/72/NCT03474172/Prot_SAP_000.pdf